CLINICAL TRIAL: NCT00770250
Title: A Mirror Assessment of the Words Used By Patients and Physicians to Express Asthma Symptoms, According To the Patient's Level of Asthma Control In General Medicine
Brief Title: National Survey on Asthma
Acronym: SYMPTOMES
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-RFR-DUM-2008/1
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Asthma
Keywords: asthma symptoms; words used by patients and physicians; express asthma symptoms
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the concordance of the most frequently used words by the patients and the physicians to express asthma symptoms, according to the patient's level of asthma control.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of persistent asthma treated with an inhaled corticosteroid based maintenance treatment for more than 3 months
* Given his/her consent to participate to the study and who is able to answer the questionnaire in french by him/her-self.

Exclusion Criteria:

* Patient with a cardiac disease (congestive heart failure, coronary artery disease)
* Patient with a respiratory disease other than asthma (COPD, sleep apnea syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first 2 consecutive patients seen during the GP's visit with a diagnosis of persistent asthma
Sampling Method: Probability Sample
Enrollment: 1704 (Actual)
Dates: Start 2008-09; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The concordance of the most frequently used words by the patients and the physicians to express asthma symptoms, according to the patient's level of asthma control. | Once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Study Director — AstraZeneca
Locations (905):
- France (905):
  - Research Site, Abbeville
  - Research Site, Ablon-sur-Seine
  - Research Site, Agneaux
  - Research Site, Agon-Coutainville
  - Research Site, Aignay-le-Duc
  - Research Site, Aigrefeuille-d'Aunis
  - Research Site, Aigrefeuille-sur-Maine
  - Research Site, Aigurande
  - Research Site, Airvault
  - Research Site, Aiserey
  - Research Site, Aix-en-Provence
  - Research Site, Ajaccio
  - Research Site, Alès
  - Research Site, Alligny-Cosne
  - Research Site, Allonnes
  - Research Site, Althen-des-Paluds
  - Research Site, Ambazac
  - Research Site, Ambès
  - Research Site, Amiens
  - Research Site, Andé
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Angers
  - Research Site, Anglet
  - Research Site, Angoulême
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Anzin
  - Research Site, Argences
  - Research Site, Argenteuil
  - Research Site, Arques-la-Bataille
  - Research Site, Arsac
  - Research Site, Arudy
  - Research Site, Aspiran
  - Research Site, Athis-Mons
  - Research Site, Aubenas
  - Research Site, Auchel
  - Research Site, Audierne
  - Research Site, Audincourt
  - Research Site, Aulnay-sous-Bois
  - Research Site, Auriol
  - Research Site, Autrans
  - Research Site, Autun
  - Research Site, Auvers-sur-Oise
  - Research Site, Auxi-le-Château
  - Research Site, Auxonne
  - Research Site, Avelin
  - Research Site, Avignon
  - Research Site, Axat
  - Research Site, Bagneux
  - Research Site, Bagnères-de-Bigorre
  - Research Site, Bagnolet
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baignes Ste Radegonde
  - Research Site, Baillet-en-France
  - Research Site, Balaruc-le-Vieux
  - Research Site, Ballon
  - Research Site, Balma
  - Research Site, Barentin
  - Research Site, Basse-Goulaine
  - Research Site, Bassillac
  - Research Site, Bayonne
  - Research Site, Bâgé-le-Châtel
  - Research Site, Beaulieu-sur-Dordogne
  - Research Site, Beaumetz-lès-Aire
  - Research Site, Beaumont
  - Research Site, Beaumont-sur-Oise
  - Research Site, Bellac
  - Research Site, Bellegarde-sur-Valserine
  - Research Site, Belleville-sur-Meuse
  - Research Site, Bellême
  - Research Site, Bergerac
  - Research Site, Bergues
  - Research Site, Berre-l'Étang
  - Research Site, Bersée
  - Research Site, Beuvrages
  - Research Site, Bezons
  - Research Site, Béziers
  - Research Site, Biganos
  - Research Site, Bihorel
  - Research Site, Billy-Montigny
  - Research Site, Blangy-sur-Bresle
  - Research Site, Blénod-lès-Pont-à-Mousson
  - Research Site, Blotzheim
  - Research Site, Boën-sur-Lignon
  - Research Site, Bohars
  - Research Site, Boos
  - Research Site, Bordeaux
  - Research Site, Bords
  - Research Site, Bormes-les-Mimosas
  - Research Site, Bort-les-Orgues
  - Research Site, Bouère
  - Research Site, Bouffémont
  - Research Site, Bougival
  - Research Site, Bourbriac
  - Research Site, Bourg-Achard
  - Research Site, Bourg-la-Reine
  - Research Site, Bourron-Marlotte
  - Research Site, Bourth
  - Research Site, Bousbecque
  - Research Site, Bouzonville
  - Research Site, Boynes
  - Research Site, Brax
  - Research Site, Brebières
  - Research Site, Brest
  - Research Site, Breuil-le-Sec
  - Research Site, Brignoud
  - Research Site, Broût-Vernet
  - Research Site, Bruay-la-Buissière
  - Research Site, Bucquoy
  - Research Site, Bulgnéville
  - Research Site, Bussang
  - Research Site, Bussy-Saint-Georges
  - Research Site, Calvisson
  - Research Site, Canet-en-Roussillon
  - Research Site, Cannes
  - Research Site, Canteleu
  - Research Site, Cany-Barville
  - Research Site, Capdenac-Gare
  - Research Site, Capestang
  - Research Site, Carbon-Blanc
  - Research Site, Carcassonne
  - Research Site, Carhaix-Plouguer
  - Research Site, Carresse-Cassaber
  - Research Site, Carvin
  - Research Site, Cassis
  - Research Site, Castelnau-Montratier
  - Research Site, Castres
  - Research Site, Caudebec-lès-Elbeuf
  - Research Site, Caulnes
  - Research Site, Caylus
  - Research Site, Cernay
  - Research Site, Cénac
  - Research Site, Cérilly
  - Research Site, Chacé
  - Research Site, Chalais
  - Research Site, Chaleins
  - Research Site, Chalindrey
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambly
  - Research Site, Champagné-les-Marais
  - Research Site, Champagnole
  - Research Site, Champeix
  - Research Site, Champigny-sur-Marne
  - Research Site, Champniers
  - Research Site, Chanceaux-sur-Choisille
  - Research Site, Chantonnay
  - Research Site, Chaource
  - Research Site, Charensat
  - Research Site, Charenton-le-Pont
  - Research Site, Charleville-Mézières
  - Research Site, Charroux
  - Research Site, Chauvigny
  - Research Site, Chavanges
  - Research Site, Chazay-d'Azergues
  - Research Site, Châlons-en-Champagne
  - Research Site, Château-d'Olonne
  - Research Site, Château-Thierry
  - Research Site, Châteaubriant
  - Research Site, Châteaugay
  - Research Site, Châteauneuf-sur-Cher
  - Research Site, Châteauroux
  - Research Site, Châtenay-Malabry
  - Research Site, Châtenois
  - Research Site, Châtillon-en-Vendelais
  - Research Site, Châtillon-sur-Chalaronne
  - Research Site, Cherbourg Octeville
  - Research Site, Choisey
  - Research Site, Choisy-le-Roi
  - Research Site, Cholet
  - Research Site, Ciboure
  - Research Site, Cires-lès-Mello
  - Research Site, Civrac-de-Blaye
  - Research Site, Clairac
  - Research Site, Clamart
  - Research Site, Clapiers
  - Research Site, Clermont-Ferrand
  - Research Site, Clessé
  - Research Site, Cognac
  - Research Site, Colleville-Montgomery
  - Research Site, Colmar
  - Research Site, Colomars
  - Research Site, Colombey-les-Belles
  - Research Site, Colomiers
  - Research Site, Combs-la-Ville
  - Research Site, Conches-sur-Gondoire
  - Research Site, Condé-sur-Noireau
  - Research Site, Conflans Ste Honorine
  - Research Site, Corbeil-Essonnes
  - Research Site, Corné
  - Research Site, Corsept
  - Research Site, Corseul
  - Research Site, Coudekerque-Branche
  - Research Site, Courbevoie
  - Research Site, Courcelles-lès-Lens
  - Research Site, Courçon
  - Research Site, Cournon-d'Auvergne
  - Research Site, Courpière
  - Research Site, Coursan
  - Research Site, Courtry
  - Research Site, Couze-et-Saint-Front
  - Research Site, Creil
  - Research Site, Créteil
  - Research Site, Criquetot-l'Esneval
  - Research Site, Crolles
  - Research Site, Cros-de-Cagnes
  - Research Site, Cugnaux
  - Research Site, Cysoing
  - Research Site, Dangé-Saint-Romain
  - Research Site, Danjoutin
  - Research Site, Deûlémont
  - Research Site, Décines-Charpieu
  - Research Site, Dieuze
  - Research Site, Diéval
  - Research Site, Digne-les-Bains
  - Research Site, Digoin
  - Research Site, Dijon
  - Research Site, Docelles
  - Research Site, Dole
  - Research Site, Douarnenez
  - Research Site, Douchy-les-Mines
  - Research Site, Dourdan
  - Research Site, Drancy
  - Research Site, Drap
  - Research Site, Dun-le-Palestel
  - Research Site, Dunkirk
  - Research Site, Eaubonne
  - Research Site, Elna
  - Research Site, Enveig
  - Research Site, Ermont
  - Research Site, Esquerdes
  - Research Site, Essars
  - Research Site, Essey-lès-Nancy
  - Research Site, Excideuil
  - Research Site, Exincourt
  - Research Site, Échirolles
  - Research Site, Élancourt
  - Research Site, Épernay
  - Research Site, Épieds-en-Beauce
  - Research Site, Épinay-sur-Seine
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Étain
  - Research Site, Étampes
  - Research Site, Étival-Clairefontaine
  - Research Site, Étupes
  - Research Site, Évaux-les-Bains
  - Research Site, Évin-Malmaison
  - Research Site, Évry
  - Research Site, Falaise
  - Research Site, Feignies
  - Research Site, Fenain
  - Research Site, Fermanville
  - Research Site, Feurs
  - Research Site, Fécamp
  - Research Site, Firminy
  - Research Site, Fitilieu
  - Research Site, Fleurance
  - Research Site, Fleury-les-Aubrais
  - Research Site, Fleury-sur-Andelle
  - Research Site, Fleury-sur-Orne
  - Research Site, Florac
  - Research Site, Folembray
  - Research Site, Fontaine
  - Research Site, Fontenay-sous-Bois
  - Research Site, Forges-les-Eaux
  - Research Site, Fos-sur-Mer
  - Research Site, Fougères
  - Research Site, Foussais-Payré
  - Research Site, Franconville
  - Research Site, Fronton
  - Research Site, Fumay
  - Research Site, Gagny
  - Research Site, Gaillefontaine
  - Research Site, Gallardon
  - Research Site, Gandrange
  - Research Site, Gap
  - Research Site, Gauchy
  - Research Site, Gelles
  - Research Site, Gelos
  - Research Site, Gennevilliers
  - Research Site, Gentilly
  - Research Site, Ger
  - Research Site, Gerbéviller
  - Research Site, Gerzat
  - Research Site, Gif-sur-Yvette
  - Research Site, Givors
  - Research Site, Gondrecourt-le-Château
  - Research Site, Gondreville
  - Research Site, Gorges
  - Research Site, Goudelin
  - Research Site, Grand-Couronne
  - Research Site, Granville
  - Research Site, Graulhet
  - Research Site, Grenade
  - Research Site, Grenoble
  - Research Site, Gréoux-les-Bains
  - Research Site, Grignols
  - Research Site, Guenrouet
  - Research Site, Guerlesquin
  - Research Site, Guichen
  - Research Site, Guidel
  - Research Site, Guingamp
  - Research Site, Guiscriff
  - Research Site, Guise
  - Research Site, Guînes
  - Research Site, Guîtres
  - Research Site, Gy
  - Research Site, Hallennes-lez-Haubourdin
  - Research Site, Halluin
  - Research Site, Hatten
  - Research Site, Haubourdin
  - Research Site, Hazebrouck
  - Research Site, Hede
  - Research Site, Hendaye
  - Research Site, Henrichemont
  - Research Site, Herbault
  - Research Site, Herblay-sur-Seine
  - Research Site, Hermonville
  - Research Site, Heyrieux
  - Research Site, Hillion
  - Research Site, Hirson
  - Research Site, Houplin-Ancoisne
  - Research Site, Hourtin
  - Research Site, Houtaud
  - Research Site, Huriel
  - Research Site, Hyères
  - Research Site, Hœrdt
  - Research Site, Igé
  - Research Site, Illiers-Combray
  - Research Site, Inguiniel
  - Research Site, Issé
  - Research Site, Issoire
  - Research Site, Issy-les-Moulineaux
  - Research Site, Istres
  - Research Site, Ivry-sur-Seine
  - Research Site, Jacou
  - Research Site, Jardin
  - Research Site, Jargeau
  - Research Site, Jeumont
  - Research Site, Jonquières-Saint-Vincent
  - Research Site, Jouars-Pontchartrain
  - Research Site, Joué-lès-Tours
  - Research Site, Juan-les-Pins
  - Research Site, Jugon-les-Lacs
  - Research Site, Jussey
  - Research Site, Juvigné
  - Research Site, Jœuf
  - Research Site, Kernilis
  - Research Site, L'Aigle
  - Research Site, L'Escarène
  - Research Site, L'Isle-Jourdain
  - Research Site, L'Isle-sur-la-Sorgue
  - Research Site, L'Île-Saint-Denis
  - Research Site, La Chaise-Dieu
  - Research Site, La Colle-sur-Loup
  - Research Site, La Ferté-Saint-Aubin
  - Research Site, La Garde
  - Research Site, La Garnache
  - Research Site, La Haye-du-Puits
  - Research Site, La Haye-Pesnel
  - Research Site, La Madeleine
  - Research Site, La Mailleraye-sur-Seine
  - Research Site, La Mure
  - Research Site, La Neuville-Roy
  - Research Site, La Riche
  - Research Site, La Roche-en-Brenil
  - Research Site, La Roche-sur-Foron
  - Research Site, La Sauve
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Teste-de-Buch
  - Research Site, La Trinité-sur-Mer
  - Research Site, La Tronche
  - Research Site, Labarthe-sur-Lèze
  - Research Site, Labenne
  - Research Site, Lachapelle-aux-Pots
  - Research Site, Lagarde-Enval
  - Research Site, Lailly-en-Val
  - Research Site, Laissac
  - Research Site, Lamagistère
  - Research Site, Lamalou-les-Bains
  - Research Site, Lamballe
  - Research Site, Lambersart
  - Research Site, Lamorlaye
  - Research Site, Landemont
  - Research Site, Landes
  - Research Site, Landouge
  - Research Site, Langres
  - Research Site, Lanouaille
  - Research Site, Lans
  - Research Site, Larmor-Baden
  - Research Site, Larmor-Plage
  - Research Site, Lasseube
  - Research Site, Lathus-Saint-Rémy
  - Research Site, Lattes
  - Research Site, Laudun-lArdoise
  - Research Site, Laure
  - Research Site, Laval
  - Research Site, Le Barcarès
  - Research Site, Le Blanc-Mesnil
  - Research Site, Le Cailar
  - Research Site, Le Cannet
  - Research Site, Le Cendre
  - Research Site, Le Coudray-Montceaux
  - Research Site, Le Fenouiller
  - Research Site, Le Fleix
  - Research Site, Le Golfe Juan
  - Research Site, Le Havre
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Lavandou
  - Research Site, Le Louroux Béconnais
  - Research Site, Le Mans
  - Research Site, Le Mesnil-Esnard
  - Research Site, Le Neubourg
  - Research Site, Le Perray-en-Yvelines
  - Research Site, Le Perréon
  - Research Site, Le Pertre
  - Research Site, Le Plessis-Trévise
  - Research Site, Le Pradet
  - Research Site, Le Pré-Saint-Gervais
  - Research Site, Le Puy-en-Velay
  - Research Site, Le Raincy
  - Research Site, Le Teil
  - Research Site, Le Touquet-Paris-Plage
  - Research Site, Le Veurdre
  - Research Site, Le Vigan
  - Research Site, Lembach
  - Research Site, Lens
  - Research Site, Les Forges
  - Research Site, Les Hautes-Rivières
  - Research Site, Les Issambres
  - Research Site, Les Lilas
  - Research Site, Les Mées
  - Research Site, Les Milles
  - Research Site, Les Pujols
  - Research Site, Les Sables-d'Olonne
  - Research Site, Lesconil
  - Research Site, Levallois-Perret
  - Research Site, Lherm
  - Research Site, Liévin
  - Research Site, Lignan-sur-Orb
  - Research Site, Lille
  - Research Site, Limeil-Brévannes
  - Research Site, Limogne-en-Quercy
  - Research Site, Linas
  - Research Site, Lingolsheim
  - Research Site, Lisses
  - Research Site, Loison-sous-Lens
  - Research Site, Longages
  - Research Site, Longpont-sur-Orge
  - Research Site, Longueau
  - Research Site, Longué-Jumelles
  - Research Site, Lons-le-Saunier
  - Research Site, Loos-en-Gohelle
  - Research Site, Lorient
  - Research Site, Lourdes
  - Research Site, Louvigné-du-Désert
  - Research Site, Lumes
  - Research Site, Lunéville
  - Research Site, Lurcy-Lévis
  - Research Site, Luxé
  - Research Site, Lyon
  - Research Site, Maignelay-Montigny
  - Research Site, Maintenon
  - Research Site, Mainvilliers
  - Research Site, Maisons-Laffitte
  - Research Site, Malaucène
  - Research Site, Malemort-sur-Corrèze
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Manduel
  - Research Site, Manosque
  - Research Site, Mantes-la-Jolie
  - Research Site, Marle
  - Research Site, Marlenheim
  - Research Site, Marsannay-la-Côte
  - Research Site, Marseille
  - Research Site, Martigues
  - Research Site, Martinvast
  - Research Site, Masevaux
  - Research Site, Masseret
  - Research Site, Matha
  - Research Site, Mauléon-Licharre
  - Research Site, Maurepas
  - Research Site, Mazan
  - Research Site, Meaulne
  - Research Site, Melle
  - Research Site, Mennevret
  - Research Site, Merkwiller-Pechelbronn
  - Research Site, Merlimont
  - Research Site, Merville
  - Research Site, Metz
  - Research Site, Meulan-en-Yvelines
  - Research Site, Meylan
  - Research Site, Mezel
  - Research Site, Mezzavia
  - Research Site, Méréville
  - Research Site, Mérignac
  - Research Site, Mézidon-Canon
  - Research Site, Mézilles
  - Research Site, Migennes
  - Research Site, Milhaud
  - Research Site, Mions
  - Research Site, Miramont-de-Guyenne
  - Research Site, Mirebeau-sur-Bèze
  - Research Site, Mirecourt
  - Research Site, Moirans
  - Research Site, Moissac
  - Research Site, Moncontour de Bretagne
  - Research Site, Monestier-de-Clermont
  - Research Site, Monéteau
  - Research Site, Mont-de-Marsan
  - Research Site, Montauban
  - Research Site, Montbazens
  - Research Site, Montbenoît
  - Research Site, Montbron
  - Research Site, Montceau-les-Mines
  - Research Site, Montcy-Notre-Dame
  - Research Site, Montebourg
  - Research Site, Montereau-Fault-Yonne
  - Research Site, Monteux
  - Research Site, Montfavet
  - Research Site, Montguyon
  - Research Site, Montigny-lès-Cormeilles
  - Research Site, Montigny-lès-Metz
  - Research Site, Montlouis-sur-Loire
  - Research Site, Montluçon
  - Research Site, Montmagny
  - Research Site, Montmain
  - Research Site, Montmorillon
  - Research Site, Montoir-de-Bretagne
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montreuil-Juigné
  - Research Site, Montrond-les-Bains
  - Research Site, Morangis
  - Research Site, Morsang-sur-Orge
  - Research Site, Mouchin
  - Research Site, Mouilleron-le-Captif
  - Research Site, Mourioux-Vieilleville
  - Research Site, Mourmelon-le-Petit
  - Research Site, Moutiers-les-Mauxfaits
  - Research Site, Mulhouse
  - Research Site, Nancy
  - Research Site, Nangis
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Nanteuil-en-Vallée
  - Research Site, Narbonne
  - Research Site, Neauphle-le-Château
  - Research Site, Nemours
  - Research Site, Neufchâtel-en-Bray
  - Research Site, Neuville-sur-Saône
  - Research Site, Nevers
  - Research Site, Nexon
  - Research Site, Nègrepelisse
  - Research Site, Nice
  - Research Site, Niederschaeffolsheim
  - Research Site, Nieppe
  - Research Site, Nieuil-l'Espoir
  - Research Site, Nîmes
  - Research Site, Nogent-le-Phaye
  - Research Site, Nogent-le-Rotrou
  - Research Site, Noirmoutier-en-l'Île
  - Research Site, Noisy-le-Grand
  - Research Site, Nordausques
  - Research Site, Nortkerque
  - Research Site, Notre-Dame-de-Monts
  - Research Site, Nouan-le-Fuzelier
  - Research Site, Nouâtre
  - Research Site, Noyelles-sous-Lens
  - Research Site, Nœux-les-Mines
  - Research Site, Obernai
  - Research Site, Oermingen
  - Research Site, Oignies
  - Research Site, Oisemont
  - Research Site, Ondres
  - Research Site, Oradour-sur-Vayres
  - Research Site, Orbey
  - Research Site, Orchamps
  - Research Site, Orchies
  - Research Site, Orgères
  - Research Site, Orly
  - Research Site, Orry-la-Ville
  - Research Site, Orvault
  - Research Site, Ouroux-sur-Saône
  - Research Site, Paillencourt
  - Research Site, Paimpont
  - Research Site, Parcey
  - Research Site, Pardies
  - Research Site, Parigné-l'Évêque
  - Research Site, Paris
  - Research Site, Parthenay
  - Research Site, Pau
  - Research Site, Peltre
  - Research Site, Penmarch
  - Research Site, Pernes-les-Fontaines
  - Research Site, Perpignan
  - Research Site, Perros-Guirec
  - Research Site, Persac
  - Research Site, Pertuis
  - Research Site, Petit-Couronne
  - Research Site, Périgueux
  - Research Site, Pézenas
  - Research Site, Pibrac
  - Research Site, Pignans
  - Research Site, Pins-Justaret
  - Research Site, Pinsaguel
  - Research Site, Pithiviers
  - Research Site, Plabennec
  - Research Site, Plaisance-du-Touch
  - Research Site, Plérin
  - Research Site, Ploeren
  - Research Site, Plonévez-du-Faou
  - Research Site, Plourhan
  - Research Site, Plourin-lès-Morlaix
  - Research Site, Plouzané
  - Research Site, Pocé-sur-Cisse
  - Research Site, Poissy
  - Research Site, Poligny
  - Research Site, Poncin
  - Research Site, Pont de Briques Saint Etienne
  - Research Site, Pont-à-Mousson
  - Research Site, Pont-de-l'Arche
  - Research Site, Pont-de-Veyle
  - Research Site, Pont-Évêque
  - Research Site, Pont-Remy
  - Research Site, Pont-Scorff
  - Research Site, Pontault-Combault
  - Research Site, Pontrieux
  - Research Site, Pornic
  - Research Site, Port Leucate
  - Research Site, Port-de-Bouc
  - Research Site, Pouzay
  - Research Site, Pradines
  - Research Site, Préchac
  - Research Site, Privas
  - Research Site, Prix-lès-Mézières
  - Research Site, Provins
  - Research Site, Puget-Ville
  - Research Site, Pulnoy
  - Research Site, Quarante
  - Research Site, Quiberon
  - Research Site, Quimper
  - Research Site, Rabastens-de-Bigorre
  - Research Site, Raismes
  - Research Site, Rambervillers
  - Research Site, Ramonville-Saint-Agne
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Restigné
  - Research Site, Rethel
  - Research Site, Rezé
  - Research Site, Réding
  - Research Site, Ribécourt-Dreslincourt
  - Research Site, Rieumes
  - Research Site, Rieux
  - Research Site, Rigney
  - Research Site, Rilhac-Rancon
  - Research Site, Rion-des-Landes
  - Research Site, Riquewihr
  - Research Site, Rivery
  - Research Site, Rixheim
  - Research Site, Roanne
  - Research Site, Robion
  - Research Site, Roche-la-Molière
  - Research Site, Roche-lez-Beaupré
  - Research Site, Rohrbach-lès-Bitche
  - Research Site, Roissy-en-France
  - Research Site, Romagnat
  - Research Site, Rombas
  - Research Site, Romorantin-Lanthenay
  - Research Site, Rosières-en-Santerre
  - Research Site, Rosny-sous-Bois
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rougegoutte
  - Research Site, Rouillac
  - Research Site, Roulans
  - Research Site, Routot
  - Research Site, Rouxmesnil-Bouteilles
  - Research Site, Rueil-Malmaison
  - Research Site, Ruelisheim
  - Research Site, Ruynes-en-Margeride
  - Research Site, Saâcy-sur-Marne
  - Research Site, Saffré
  - Research Site, Sains-du-Nord
  - Research Site, Saint Georges Baillargeaux
  - Research Site, Saint-Affrique
  - Research Site, Saint-Aigulin
  - Research Site, Saint-Amand-Montrond
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Anthème
  - Research Site, Saint-Antonin-Noble-Val
  - Research Site, Saint-Arnoult-en-Yvelines
  - Research Site, Saint-Astier
  - Research Site, Saint-Aubert
  - Research Site, Saint-Aunès
  - Research Site, Saint-Avold
  - Research Site, Saint-Branchs
  - Research Site, Saint-Brevin-les-Pins
  - Research Site, Saint-Chaffrey
  - Research Site, Saint-Christol-les-Alès
  - Research Site, Saint-Claude-de-Diray
  - Research Site, Saint-Cyprien
  - Research Site, Saint-Cyr-sur-Mer
  - Research Site, Saint-Denis
  - Research Site, Saint-Dizier
  - Research Site, Saint-Etienne
  - Research Site, Saint-Etienne-de-Tulmont
  - Research Site, Saint-Égrève
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Étienne-de-Saint-Geoirs
  - Research Site, Saint-Étienne-du-Rouvray
  - Research Site, Saint-Évarzec
  - Research Site, Saint-Fargeau-Ponthierry
  - Research Site, Saint-Féliu-d'Avall
  - Research Site, Saint-Geniès-de-Malgoirès
  - Research Site, Saint-Genis-les-Ollières
  - Research Site, Saint-Georges-dOrques
  - Research Site, Saint-Germain-Lembron
  - Research Site, Saint-Germain-sur-Morin
  - Research Site, Saint-Gervais-en-Belin
  - Research Site, Saint-Gratien
  - Research Site, Saint-Hilaire-du-Harcouët
  - Research Site, Saint-Jean-de-la-Ruelle
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-de-Monts
  - Research Site, Saint-Jean-le-Blanc
  - Research Site, Saint-Jeannet
  - Research Site, Saint-Just-en-Chaussée
  - Research Site, Saint-Lambert-la-Potherie
  - Research Site, Saint-Laurent-Blangy
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Laurent-en-Caux
  - Research Site, Saint-Léger-des-Vignes
  - Research Site, Saint-Léger-lès-Domart
  - Research Site, Saint-Léonard-de-Noblat
  - Research Site, Saint-Marcellin
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-du-Var
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Médard-en-Jalles
  - Research Site, Saint-Michel-en-lHerm
  - Research Site, Saint-Omer
  - Research Site, Saint-Palais-sur-Mer
  - Research Site, Saint-Philbert-de-Bouaine
  - Research Site, Saint-Pierre-de-Fursac
  - Research Site, Saint-Pol-sur-Ternoise
  - Research Site, Saint-Pourçain-sur-Sioule
  - Research Site, Saint-Priest
  - Research Site, Saint-Quentin
  - Research Site, Saint-Rambert-d'Albon
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Rémy-la-Varenne
  - Research Site, Saint-Rome-de-Cernon
  - Research Site, Saint-Saëns
  - Research Site, Saint-Savinien
  - Research Site, Saint-Savournin
  - Research Site, Saint-Sever
  - Research Site, Saint-Sébastien-sur-Loire
  - Research Site, Saint-Sylvain
  - Research Site, Saint-Thuriau
  - Research Site, Saint-Vallier
  - Research Site, Saint-Yorre
  - Research Site, Saintes
  - Research Site, Salbris
  - Research Site, Salomé
  - Research Site, Sanary-sur-Mer
  - Research Site, Saran
  - Research Site, Sarre-Union
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Sassenage
  - Research Site, Saulnot
  - Research Site, Saulon-la-Chapelle
  - Research Site, Sault-lès-Rethel
  - Research Site, Saulxures-lès-Nancy
  - Research Site, Savigny-le-Temple
  - Research Site, Savonnières
  - Research Site, Schiltigheim
  - Research Site, Seclin
  - Research Site, Sedan
  - Research Site, Segré
  - Research Site, Semblançay
  - Research Site, Sens
  - Research Site, Sens-de-Bretagne
  - Research Site, Sentheim
  - Research Site, Sepmeries
  - Research Site, Septèmes-les-Vallons
  - Research Site, Sequedin
  - Research Site, Seraincourt
  - Research Site, Seysses
  - Research Site, Sète
  - Research Site, Sierck-les-Bains
  - Research Site, Simiane-Collongue
  - Research Site, Six-Fours-les-Plages
  - Research Site, Socx
  - Research Site, Soissons
  - Research Site, Soisy-sous-Montmorency
  - Research Site, Solesmes
  - Research Site, Solliès-Pont
  - Research Site, Somain
  - Research Site, Sonchamp
  - Research Site, Soufflenheim
  - Research Site, Soyaux
  - Research Site, St-Malo
  - Research Site, Stains
  - Research Site, Ste Florine
  - Research Site, Ste Fortunade
  - Research Site, Ste Foy de Peyrolieres
  - Research Site, Ste Severe Sur Indre
  - Research Site, Strasbourg
  - Research Site, Sucy-en-Brie
  - Research Site, Tabanac
  - Research Site, Tarascon
  - Research Site, Tarbes
  - Research Site, Tarcenay
  - Research Site, Tartas
  - Research Site, Tencin
  - Research Site, Tessy-sur-Vire
  - Research Site, Thilouze
  - Research Site, Thionville
  - Research Site, Thonon-les-Bains
  - Research Site, Thuir
  - Research Site, Thuré
  - Research Site, Til-Châtel
  - Research Site, Tincques
  - Research Site, Tonneins
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tournan-en-Brie
  - Research Site, Tours
  - Research Site, Toussieu
  - Research Site, Tracy-le-Mont
  - Research Site, Traînel
  - Research Site, Trets
  - Research Site, Trélissac
  - Research Site, Trieux
  - Research Site, Trith-Saint-Léger
  - Research Site, Truchtersheim
  - Research Site, Tulette
  - Research Site, Tulle
  - Research Site, Uchaud
  - Research Site, Uzès
  - Research Site, Vailly-sur-Aisne
  - Research Site, Vaison-la-Romaine
  - Research Site, Valenciennes
  - Research Site, Vanault-les-Dames
  - Research Site, Varangéville
  - Research Site, Vatan
  - Research Site, Vaugneray
  - Research Site, Vaulx-en-Velin
  - Research Site, Veigné
  - Research Site, Vendenheim
  - Research Site, Vendôme
  - Research Site, Vennecy
  - Research Site, Verdun
  - Research Site, Vern-sur-Seiche
  - Research Site, Vernet
  - Research Site, Verny
  - Research Site, Versailles
  - Research Site, Vert-Saint-Denis
  - Research Site, Vertou
  - Research Site, Vervins
  - Research Site, Vestric-et-Candiac
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vic-sur-Aisne
  - Research Site, Vichy
  - Research Site, Vieille-Église
  - Research Site, Vif
  - Research Site, Villefagnan
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villefranche-sur-Mer
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villejuif
  - Research Site, Villemomble
  - Research Site, Villeneuve les beziers
  - Research Site, Villeneuve-la-Garenne
  - Research Site, Villeneuve-lès-Avignon
  - Research Site, Villeneuve-Loubet
  - Research Site, Villeneuve-Tolosane
  - Research Site, Villenoy
  - Research Site, Villeparisis
  - Research Site, Villeurbanne
  - Research Site, Villiers-le-Bel
  - Research Site, Virieu Sur Bourbre
  - Research Site, Viry-Châtillon
  - Research Site, Vitré
  - Research Site, Vitrolles
  - Research Site, Vitry-sur-Seine
  - Research Site, Viviers
  - Research Site, Voiron
  - Research Site, Vouillé
  - Research Site, Voujeaucourt
  - Research Site, Vouziers
  - Research Site, Wambrechies
  - Research Site, Wasselonne
  - Research Site, Wattrelos
  - Research Site, Westhoffen
  - Research Site, Wissembourg
  - Research Site, Woippy
  - Research Site, Yerville
  - Research Site, Yffiniac
  - Research Site, Zuydcoote